CLINICAL TRIAL: NCT00058435
Title: Phase I Trial of the Monoclonal Anti-Idiotype Antibody ACA125 in Patients With Epithelial Ovarian, Fallopian Tube, or Peritoneal Cancer
Brief Title: Monoclonal Antibody Vaccine Therapy in Treating Patients With Ovarian Epithelial, Fallopian Tube, or Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 02-122; CDR0000288831 (Registry Identifier: PDQ (Physician Data Query)); CELLCONTROL-MSKCC-02122
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — abagovomab

INTERVENTIONS:
Biological: abagovomab

SUMMARY:
RATIONALE: Vaccines made from monoclonal antibodies combined with tumor cells may make the body build an immune response to kill tumor cells.

PURPOSE: Randomized phase I trial to study the effectiveness of vaccine therapy in treating patients who have ovarian epithelial, fallopian tube, or peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of varying routes and doses of monoclonal antibody ACA125 anti-idiotype vaccine in patients with ovarian epithelial, fallopian tube, or peritoneal cancer.
* Determine an optimal dose and route of this vaccine for a phase II study.
* Determine the immune response induced by this vaccination in these patients.
* Determine the time to development of objective tumor response in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive lower-dose monoclonal antibody ACA125 anti-idiotype vaccine (MOAB ACA125) intramuscularly (IM) on weeks 0, 2, 4, 6, 10, and 14 in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive higher-dose MOAB ACA125 IM as in arm I.
* Arm III: Patients receive lower-dose MOAB ACA125 subcutaneously (SC) on weeks 0, 2, 4, 6, 10, and 14 in the absence of disease progression or unacceptable toxicity.
* Arm IV: Patients receive higher-dose MOAB ACA125 SC as in arm III. Patients are followed every 6-12 weeks for 2 years.

PROJECTED ACCRUAL: A total of 40 patients (10 patients per cohort) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, fallopian tube, or peritoneal cancer

  * Stage II-IV
* Initially treated with surgery and at least 1 platinum-based chemotherapy regimen
* Must have relapsed after initial treatment and completed chemotherapy for recurrent disease
* Asymptomatic residual measurable disease on CT scan and/or an elevated CA 125 allowed
* Complete clinical remission allowed, defined by the following criteria:

  * CA 125 no greater than 35 IU/mL
  * No objective evidence of disease by CT scan
  * Normal physical examination

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* At least 3 months

Hematopoietic

* WBC at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin no greater than 2 times normal
* ALT no greater than 2 times normal
* Alkaline phosphatase no greater than 2 times normal

Renal

* Creatinine no greater than 1.5 times normal

Other

* Not pregnant or nursing
* No potential for child bearing
* Human antimurine antibody negative
* HIV negative
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No active infection
* No known autoimmune disease (e.g., rheumatoid arthritis or ulcerative colitis)
* No known immune deficiency (e.g., hypogammaglobulinemia)
* No known allergy to murine proteins

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 6 weeks since prior interferon
* At least 6 weeks since prior immunotherapy or biological response modifiers
* No prior anticancer vaccine

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior cytotoxic or investigational chemotherapy

Endocrine therapy

* No concurrent steroids

Radiotherapy

* At least 4 weeks since prior radiotherapy

Surgery

* See Disease Characteristics

Other

* At least 1 week since prior antibiotics
* No concurrent cyclosporine
* No other concurrent immunosuppressive therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-12; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sabbatini, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States